CLINICAL TRIAL: NCT02186574
Title: A Multi-centre Phase III Study to Evaluate Pre-emptive Tenofovir for Prevention of Hepatitis B Virus Reactivation in HBsAg Negative/Anti-HBc Positive Individuals Undergoing Anti-CD20-based Chemotherapy for Non-Hodgkin's Lymphoma or Chronic Lymphocytic Leukemia/Small Lymphocytic Leukemia
Brief Title: Tenofovir to Prevent HBV Reactivation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JF62014
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Hepatitis B; Lymphoma; Non-Hodgkin
Keywords: Non-Hodgkin; Lymphoma; Hepatitis B; Tenofovir; Viread
MeSH Terms: conditions — Hepatitis B; Lymphoma | interventions — Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-emptive tenofovir (Active Comparator): Tenofovir disoproxil
  Interventions: Drug: Tenofovir disoproxil
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Tenofovir disoproxil
  Other Names: Viread
  Arms: Pre-emptive tenofovir
Drug: Placebo Oral Tablet
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine how effective preemptive tenofovir therapy is in preventing the re-activation of Hepatitis B infection, in patients who are receiving rituximab-based chemotherapy for Non-Hodgkin's Lymphoma or CLL/SLL. The rate of re-activation will be compared between patients who receive preemptive tenofovir and patients who receive tenofovir as needed.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Diagnosis of non-Hodgkin's lymphoma to be treated with rituximab-based chemotherapy
3. HBsAg negative, anti-HBc positive

Exclusion Criteria:

1. Current therapy with known activity against HBV
2. Screening ALT > 10 x ULN
3. Screening ALT >2 and <10 xULN with HBV DNA > 2000 IU/mL (indicates active HBV infection despite HBsAg negative and require antiviral therapy)
4. Life expectancy < 3 months
5. HBsAg positive
6. HIV co-infection
7. Active HCV co-infection (HCV RNA positive)
8. Creatinine clearance <50 mL/min
9. Intolerance to tenofovir
10. Women of child-bearing potential unwilling to take contraception during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2015-05; Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Rate of reverse seroconversion | 12 months post-chemotherapy
  The difference in the rate of reverse seroconversion or Hepatitis B (HBV)-associated hepatitis (definition: appearance of HBsAg in the serum with or without detectable HBV DNA in a patient who was previously HBsAg-/cAb+.) between the intervention and placebo groups.

SECONDARY OUTCOMES:
Rates of HBV Reactivation | 12 months post-chemotherapy
Severe HBV-associated hepatitis | 12 months post-chemotherapy
HBV-related liver failure | 12 months post-chemotherapy
Liver-related death | 12 months post-chemotherapy
Treatment-related adverse effects (AEs) | 12 months post-chemotherapy
Time to start chemotherapy | 12 months post-chemotherapy
Chemotherapy interruption | 12 months post-chemotherapy
All-cause mortality | 12 months post-chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Harry Janssen, MD, Study Director — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Toronto General Hospital, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

REFERENCES:
- [Derived] Tabataba Vakili S, Hirode G, Zahoor A, Saunthar A, Feld JB, Hansen BE, Syeda A, Janssen HLA, Kukreti V, Kuruvilla J, Prica A, Cheung M, Buckstein R, Hicks L, Coffin CS, Street LE, Disperati P, Chan KK, Crump M, Feld JJ. Tenofovir alafenamide for prevention of HBV reactivation in HBsAg-negative, anti-HBc-positive patients undergoing rituximab-based chemotherapy: A multicenter randomized controlled trial. Hepatol Commun. 2025 Dec 3;9(12):e0859. doi: 10.1097/HC9.0000000000000859. eCollection 2025 Dec 1. PMID 41335575